CLINICAL TRIAL: NCT05968209
Title: The Impact of Probiotic Supplementation on General Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Welsh Ambulance Service NHS Trust (Unknown); Cultech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: proWEB
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Well-Being, Psychological
Keywords: Probiotic; Well-being; Absenteeism
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active group (Experimental)
  Interventions: Dietary Supplement: Lab4P

INTERVENTIONS:
Dietary Supplement: Lab4P — Multi-strain Probiotic Product: Lactobacillus acidophilus CUL-60, Lactobacillus acidophilus CUL-21, Lactobacillus plantarum CUL-66, Bifidobacterium bifidum CUL-20, Bifidobacterium animalis subsp lactis CUL-34 (total 50 billion bacteria), Vitamin D (400 IU), Vitamin C (80 mg) & Zinc (10 mg)

SUMMARY:
The health and wellbeing of any workforce is a core priority and taking steps to ensure the wellbeing of employees is an important part of everyday working life. Winter is a time of particular challenge and is linked to increased absenteeism. There is a growing awareness that probiotics (similar to the bacteria found in yogurts) can play a role in boosting general wellbeing. Probiotics are known as 'good' or 'friendly' bacteria and are living organisms that are found naturally in yogurt and fermented foods. They can be capsules, tablets or powders in sachets that are taken daily to help to keep the gut in peak condition. Everyone has trillions of bacteria in their guts living together happily and they are needed to boost our wellbeing but the stresses and strains of everyday life can often disturb their balance, probiotics can help to restore the balance. Over the winter of 2022, a small exploratory study with employees based in South Wales who were offered the opportunity to 'try out' a probiotic manufactured by Cultech Limited (a company based in Port Talbot specialising in the production of nutritional supplements). The results were very promising with significant improvements in wellbeing and reduced absenteeism among those who opted to take the product. This project is designed as a follow-up on last year's exploratory study to further assess effectiveness of the same probiotic nutritional supplement over the winter

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 60 (at the time of consent)
2. Working in an NHS healthcare setting
3. Willing to use the Trialflare app on personal phone to record data securely
4. Able to understand and communicate using the English language
5. Normal or corrected to normal vision 6 Happy to take no other probiotics during study

7. Able to continue with normal lifestyle throughout 8. Able to consent to take part in the study

Exclusion Criteria:

1. Immunodeficient
2. Taking probiotics or have taken within the last month
3. Allergic or suspected allergy to zinc

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life changes | 60 days
  Weekly questionnaires via an app containing questions relating to the participant's quality of life (i.e. mood, sleep, energy levels) over a week period
Change in Absenteeism | 60 days
  Weekly questionnaires via an app relating to any absences from work over a week period
Changes in gut symptoms and overall health | 60 days
  Weekly questionnaires via an app containing questions on the number of days participants may have experiences gut related symptoms (i.e. bloating, constipation, diarrhoea, stomach pain), and overall health (i.e. headaches, coughs, sore thorat)

SECONDARY OUTCOMES:
Feasibility of app-based probiotic studies | 60 days
  To gain an understanding of the level of interest amongst the workforce to take part in probiotic studies and use of an app to monitor well-being.
  Measured through levels of sign-up, collection of intervention and drop-out rate over the course of the trial. All which will be measured through the app

CONTACTS AND LOCATIONS:
Locations (1):
- Cwm Taf Morgannwg Health Board, Pontypridd, Mid Glamorgan, United Kingdom